CLINICAL TRIAL: NCT02360891
Title: Study of Predictive Factors of Progression of Motor Neurone Disease Prognosis and Endophenotype Biomarkers French Database Set up
Brief Title: Study of Predictive Factors of Progression of Motor Neurone Disease
Acronym: PULSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-50; 2013-A00969-36 (Other: ID RCB number, ANSM)
Record Dates: First submitted 2015-01-07; First posted 2015-02-11 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: multimodal biomarkers; prognosis; endophenotypes
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, platelets, cerebrospinal fluid,skin, muscle, brains
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients: follow up of patients with amyotrophic lateral sclerosis from the first signs to the end of the disease
  Interventions: Other: biomarkers (composite analysis)
- neurological controls: patients with other neurological disease
  Interventions: Other: biomarkers (composite analysis)
- healthy controls: age matched healthy controls
  Interventions: Other: biomarkers (composite analysis)

INTERVENTIONS:
Other: biomarkers (composite analysis) — biological, imaging, electrophysiological and anatomopathological examinations

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a complex polymorph and devastating neurodegenerative disease. Although the pathophysiological mechanisms underlying the development of ALS remain to be fully elucidated, there have been significant advances in the understanding of ALS pathogenesis, with evidence emerging of a complex interaction between genetic factors and dysfunction of vital molecular pathways. However, the numerous randomized clinical trials (RCT) for ALS have failed to generate improved drug treatments. Biomarkers able to bring prognostic value and to distinguish the different endophenotypes of this polymorphic disease could help to better select clusters of patients in order to improve the RCT outcomes. However, little progress has been made in the development of viable diagnostic, prognostic and monitoring markers. This could be explained by common shortcomings, such as relatively small sample sizes, statistically underpowered study designs, lack of disease controls and poorly characterized patient cohorts. It is yet crucial that the investigators further develop and validate ALS biomarkers and incorporate these biomarkers into the drug development pipeline for ALS.

The aim of the present study is therefore to determine the clinical, biological, imaging, and electrophysiological biomarkers of prognosis of survival without events (i.e. severe comorbidity, 24 hours of non invasive ventilation, tracheotomy). This is a prospective observational multicentric French study of a cohort of 1000 ALS patients.

This large multimodal database will be open for international fruitful scientific collaborations.

DETAILED DESCRIPTION:
This is a prospective observational multicentric French study of a cohort of 1000 ALS patients, 100 neurological controls and 200 healthy controls followed from the first signs to the end of the disease.

The aim of the present study is therefore to determine the clinical, biological, imaging, and electrophysiological biomarkers of prognosis of survival without events (i.e. severe comorbidity, 24 hours of non invasive ventilation, tracheotomy).

Secondary objectives will notably include i) the biomarkers of disease progression ii) biomarkers of diagnosis as compared with controls iii) the determination of the different endophenotypes according to the prognosis, the genetic profiles and the initial clinical presentations. Criteria of assessment will notably include detailed medical history, habitus, past and present treatments, vascular risk factors, ALSFRS-R, muscular testing, respiratory parameters including early nocturnal saturation and apneal profile, the detailed and predetermined clinical presentations, extensive cognitive and behavioral examination, extensive blood, cerebrospinal fluid, urines biological tests, genetic analyses, multiple brain and spinal MRI sequences, and electrophysiological tests (i.e. electromyogram, MUNIX, triple stimulation). Invasive tests will be optional (i.e. lumbar puncture, skin biopsies, muscular biopsies).

The large number of patients will allow in depth statistical analyses, notably to establish decisional trees (CHAID).

ELIGIBILITY:
Inclusion Criteria for ALS patients:

* Patients with suspicion of Amyotrophic lateral sclerosis
* Since the first signs (cramps fasciculation) or first deficit at the diagnosis work up
* Patient older than 18 years
* Patient able to provide informed consent

Inclusion Criteria for healthy controls:

* Subjects older than 18 years (matched population for age and sex with ALS)
* Neurological testing and examination showing no neurological disorders.
* Not having severe disease or life- functional prognosis

Inclusion Criteria for neurological controls:

* Patients having a typical neurodegenerative diseases other than ALS (Parkinson's disease, Alzheimer's disease)
* Not having severe disease or life- functional prognosis
* Patient older than 18 years (matched population for age and sex with ALS)
* Patient able to provide informed consent

Exclusion Criteria:

* Subjects younger than 18 years
* Patient unable to provide informed consent
* Having severe disease or life- functional prognosis
* Contraindications MRI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Multicentric French cohort of 1000 ALS patients, 100 neurological controls and 200 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change of biomarkers of survival | From date of randomization until the date of first documented progression , assessed up to 100 months
  The predictive value of the clinical, biological, imaging, and electrophysiological biomarkers of survival will be analyzed according to the life duration (months) without events (i.e. severe comorbidity, 24 hours of non invasive ventilation, tracheotomy)

SECONDARY OUTCOMES:
Change of biomarkers of disease progression | baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 24 months, 36 months, 48 months (average)
  The predictive value of the clinical, biological, imaging, and electrophysiological biomarkers of prognosis will be analyzed according to the rate of progression of the ALSFRS-R score
Clinical endophenotypes according to the survival duration | From date of randomization until the date of death related with ALS or tracheotomy or continuous non invasive ventilation (24 hours a day), whichever came first, assessed up to 100 months
  The determination of the different clinical, biological, radiological and electrophysiological endophenotypes (clusters of the same characteristics) according to the survival duration
Genetic endophenotypes | the date of death related with ALS or tracheotomy or continuous non invasive ventilation (24 hours a day), whichever came first, assessed up to 100 months
  the determination of the different clinical, biological, radiological and electrophysiological endophenotypes (clusters of the same characteristics) according to the according to the genetic forms (SOD1, TDP43, FUS, C9orf72,...)

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, MD, PhD, Study Chair — University Hospital, Lille
Locations (13):
- France (13):
  - CHU Pontchaillou, Angers
  - CHU Cote de Nacre, Caen
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHRU, Hôpital Salengro, Lille
  - Hôpital Dupuytren, Limoges
  - Hôpital Neurologique Pierre Wertheimer, Lyon
  - AP-HM,Hôpital de la Timone, Marseille
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital de l'Archet 1, CHU, Nice
  - Hôpital La Pitié (AP-HP), Paris
  - Centre Hospitalier, Saint-Brieuc
  - Hôpital Nord, Saint-Etienne
  - CHU Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grapperon AM, Harlay V, Boucekine M, Devos D, Rolland AS, Desnuelle C, Delmont E, Verschueren A, Attarian S. Could the motor unit number index be an early prognostic biomarker for amyotrophic lateral sclerosis? Clin Neurophysiol. 2024 Jul;163:47-55. doi: 10.1016/j.clinph.2024.04.013. Epub 2024 Apr 26. PMID 38703699
- [Derived] Le Gall L, Duddy WJ, Martinat C, Mariot V, Connolly O, Milla V, Anakor E, Ouandaogo ZG, Millecamps S, Laine J, Vijayakumar UG, Knoblach S, Raoul C, Lucas O, Loeffler JP, Bede P, Behin A, Blasco H, Bruneteau G, Del Mar Amador M, Devos D, Henriques A, Hesters A, Lacomblez L, Laforet P, Langlet T, Leblanc P, Le Forestier N, Maisonobe T, Meininger V, Robelin L, Salachas F, Stojkovic T, Querin G, Dumonceaux J, Butler Browne G, Gonzalez De Aguilar JL, Duguez S, Pradat PF. Muscle cells of sporadic amyotrophic lateral sclerosis patients secrete neurotoxic vesicles. J Cachexia Sarcopenia Muscle. 2022 Apr;13(2):1385-1402. doi: 10.1002/jcsm.12945. Epub 2022 Feb 22. PMID 35194965
- [Derived] Grolez G, Kyheng M, Lopes R, Moreau C, Timmerman K, Auger F, Kuchcinski G, Duhamel A, Jissendi-Tchofo P, Besson P, Laloux C, Petrault M, Devedjian JC, Perez T, Pradat PF, Defebvre L, Bordet R, Danel-Brunaud V, Devos D. MRI of the cervical spinal cord predicts respiratory dysfunction in ALS. Sci Rep. 2018 Jan 29;8(1):1828. doi: 10.1038/s41598-018-19938-2. PMID 29379040